CLINICAL TRIAL: NCT06615167
Title: A Single-blind (Data Analyst 1), Single-arm Design, Prospective, Multi-center Confirmatory Clinical Trial for Verifying the Efficacy and Safety of 'ALZGUARD' as a Digital Dementia Diagnostic Aid-Tool for the Diagnosis of the Major Neurocognitive Disorders According to DSM-5
Brief Title: Confirmatory Clinical Trial for Verifying the Efficacy and Safety of 'ALZGUARD' as a Digital Dementia Diagnostic Aid-Tool for the Diagnosis of the Major Neurocognitive Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HAII corp.ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: G00020
Record Dates: First submitted 2024-09-20; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Dementia; Major Neurocognitive Disorder
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: This is a single-arm, interventional clinical trial designed to evlauate the efficacy and safety of ALZGAURD, a smartphone-based digital therapeutic, in detecting dementia.
  Study type: interentional (clinical trial) Masking: Single-blind (Outcomes assessor) Intervention description: The ALZGUARD application will be used by participants to assess cognitive function. Results will be compared to clinical diagnoses made by neurologists.
  Primary Outcome: the accuracy of the ALZGUARD diagnosis, measured by Area Under the Curve.
Masking Description: In this study, there will be two data analysts involved. Analyst 1 will be responsible for analyzing the results generated by the ALZGUARD application, which are based on the ALZGUARD AI model. This analyst will assess whether each subject has dementia and the likelihood or probability of the diagnosis. Analyst 1 will be blinded to any clinical assessments or dianoses made by the neurologists.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ALZGUARD Intervention Group (Experimental): All participants wil use the ALZGAURD smartphone-based digital therapeutic(DTx) to assess cognitive function for detecting dementia.
  Interventions: Device: ALZGUARD

INTERVENTIONS:
Device: ALZGUARD — A digital therapeutic(DTx) application that uses artifical intelligence to analyze cognitive function and provide a diagnosis of dementia.

SUMMARY:
The goal of this clinical trial is to evalute the efficacy of ALZGUARD, a smartphone-based digital therapeutic(DTx), in comparison to diagnosis by medical doctors, as weel as to assess the safety of the application.

DETAILED DESCRIPTION:
The study will be conducted across multiple sites, enrolling participants aged 55 to 85 years olds.

The primary objective of the study is to compare the diagnositic accuracy of ALZGAURD against traditional diagnostic evaluactions conducted by medical professionals. The primary endpoint for efficacy will be the Area Under the Curve(AUC), which will measure the diagnostic performance of the application. This statistical metric will help determine how well ALZGUARD can identify dementia compared to standard diagnostic methods.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between 55 and 85 years old (both men and women).
* Participants must be able to understand and voluntarily agree to the purpose, content, and procedures of the clinical trial.

Exclusion Criteria:

* Participants with no literacy or illiteracy.
* Participants with an intellectual disability.
* Participants with presenting active psychiatric symptoms.
* Participants who have difficulty ALZGUARD application
* Participants who are unable to use a smartphone, unless they can use it with assistant.
* Participants with a history of suicidal ideation or suicidal complusion in the last 6 months.
* Other conditions as deemed inappropriate for study participant by the Principal Investigator(PI).

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) | up to 8 months
  The primary outcome will be the Area Under the Curve (AUC), which will assess the diagnostic accuracy of ALZGUARD by comparing its results with the clinical diagnosis made by neurologists. AUC will be calculated to determine the performance of ALZGUARD in detecting dementia.

SECONDARY OUTCOMES:
Sensitivity | up to 8 months
  The one of the secondary outcome will measure the sensitivity of ALZGUARD in detecting dementia. Sensitivity refers to the proportion of true positive cases accurately identified by ALZGUARD, compared to clinical diagnosis made by neurologists. This measure will assess the ability of ALZGUARD to correctly identiry patients who have dementia.
Specificity | up to 8 months
  Specificity refers to the proportion of true negative cases accurately identified by ALZGUARD, compared to the clinical diagnosis made by neurologists. This outcome will assess the ability of ALZGUARD to correctly identify patient who do not have dementia.

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Kangwon National University Hospital, Chuncheon, Gangwon-do
  - Ewha Womans University Mokdong Medical Center, Seoul
  - Yongin Severance Hospital, Seoul